CLINICAL TRIAL: NCT06564597
Title: Effectiveness of Activity-based Training After Myocardial Infarction: A Randomized Controlled Study
Brief Title: Activity-based Training After Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, HANDE USTA, Assistant Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-205945
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Ischemia; Activities of Daily Living
Keywords: Myocardial Ischemia; Activities of Daily Living; Metabolic Equivalent
MeSH Terms: conditions — Myocardial Ischemia | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal education and two brochure handouts (Experimental): The educational brochures are prepared to include clear, legible, realistic and up-to-date information. The context of the education includes the following topics:
  * What is myocardial infarction?
  * What are its clinical features?
  * Risk factors
  * Lifestyle changes
  * What is cardiac rehabilitation?
  * Stress and anxiety management
  * Energy conservation techniques
  * Progressive relaxation techniques
  Interventions: Other: Patient education
- Verbal education, two brochure handouts and MET-based activity planning (Experimental): The educational brochures are prepared to include clear, legible, realistic and up-to-date information. The context of the education includes the following topics:
  * What is myocardial infarction?
  * What are its clinical features?
  * Risk factors
  * Lifestyle changes
  * What is cardiac rehabilitation?
  * Return to activity and activity-based prescription (based on MET)
  * What are the abnormal responses that may occur in activities?
  * Stress and anxiety management
  * Energy conservation techniques
  * Progressive relaxation techniques
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Patient education — Patient education and counseling are offered one-on-one at the bedside during discharge and are also provided in the second week after discharge in an outpatient clinic setting.

SUMMARY:
Cardiovascular diseases cause high morbidity and mortality, resulting in disability, medical complications and comorbidities. Patients who have MI experience motor, cognitive and sensory impairments, reduced quality of life and burdened the national economy. Cardiac rehabilitation aims to optimize patients' health services, reduce physical and psychological effects and increase activity return performance. The rehabilitation process includes physical activities and patient education starting in the early stages after MI. Psychosocial support and occupational therapy can accelerate patients' recovery and return to daily activities. Since there are inadequacies in the literature on this subject, this study aims to provide an effective educational intervention for patients who have MI and to examine a safe return to activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myocardial infarction (ST elevation or non-ST elevation)
* Ejection fraction > 40%

Exclusion Criteria:

* Ejection fraction < 40%
* Presence of exercise-induced ischemia
* Presence of orthopedic or neurological disorder that will affect the current study
* Presence of pulmonary disease that will affect the current study (COPD, Asthma)
* Presence of visual impairment
* Presence of malignancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | The evaluation were completed after discharge. The exact time is post-operative 2nd week, 3th month and 6th month.
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
Katz Index of Independence in Activities of Daily Living | The evaluation were completed after discharge. The exact time is post-operative 2nd week, 3th month and 6th month.
  The Katz Index of Independence in Activities of Daily Living, commonly referred to as the Katz ADL, is the most appropriate instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently.
Lawton Brody Instrumental Activities of Daily Living Scale | The evaluation were completed after discharge. The exact time is post-operative 2nd week, 3th month and 6th month.
  The Lawton Instrumental Activities of Daily Living Scale (IADL) is an appropriate instrument to assess independent living skills. These skills are considered more complex than the basic activities of daily living as measured by the Katz Index of ADLs.

CONTACTS AND LOCATIONS:
Overall Officials: ALI KITIS, Professor, Study Chair — Pamukkale University Faculty of Physiotherapy and Rehabilitation
Locations (1):
- Pamukkale University, Merkez, Deni̇zli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham H, Prue-Owens K, Kirby J, Ramesh M. Systematic Review of Interventions Designed to Maintain or Increase Physical Activity Post-Cardiac Rehabilitation Phase II. Rehabil Process Outcome. 2020 Aug 25;9:1179572720941833. doi: 10.1177/1179572720941833. eCollection 2020. PMID 34497468
- [Result] CAIN HD, FRASHER WG Jr, STIVELMAN R. Graded activity program for safe return to self-care after myocardial infarction. JAMA. 1961 Jul 15;177:111-5. doi: 10.1001/jama.1961.03040280015005. No abstract available. PMID 13689828